CLINICAL TRIAL: NCT01107626
Title: Randomized Phase III Study of Maintenance Therapy With Bevacizumab, Pemetrexed, or a Combination of Bevacizumab and Pemetrexed Following Carboplatin, Paclitaxel and Bevacizumab for Advanced Non-Squamous NSCLC
Brief Title: Bevacizumab or Pemetrexed Disodium Alone or In Combination After Induction Therapy in Treating Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E5508; NCT01107626 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Paclitaxel; Carboplatin; Injections; Bevacizumab; Glutamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Induction then Maintenance with Bevacizumab) (Experimental): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm A receive bevacizumab IV over 30-90 minutes on day 1 of every cycle until progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Bevacizumab
- Arm B (Induction then Maintenance with Pemetrexed) (Experimental): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm B receive pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Bevacizumab; Drug: Pemetrexed Disodium Heptahydrate
- Arm C (Induction then Maintenance with Bevacizumab & Pemetrexed) (Experimental): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm C receive bevacizumab as in arm A and pemetrexed as in arm B.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Bevacizumab; Drug: Pemetrexed Disodium Heptahydrate

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Taxol; NSC 673089
Drug: Carboplatin — Given IV
  Other Names: carboplatin for injection or platinum diamine [1,1-cyclobutane-decarbozxylate (2-0,0')-,(SP-4-2)]
Biological: Bevacizumab — Given IV
  Other Names: NSC 704865; RhuMAb VEGF; Recombinant Humanized Monoclonal Anti-VEGF Antibody
Drug: Pemetrexed Disodium Heptahydrate — Given IV
  Other Names: L-Glutamic acid; N-[4-[2-(2-amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-; disodium salt; heptahydrate
  Arms: Arm B (Induction then Maintenance with Pemetrexed); Arm C (Induction then Maintenance with Bevacizumab & Pemetrexed)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Pemetrexed disodium may stop the growth of tumor cells by blocking some enzymes needed for cell growth. It is not yet known whether giving bevacizumab or pemetrexed disodium alone or in combination is more effective in treating non-squamous non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying bevacizumab and pemetrexed disodium alone or in combination after induction therapy to see how well they work in treating patients with advanced non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the overall survival (OS) of patients with advanced non-squamous non-small cell lung cancer (NSCLC) treated with maintenance therapy with bevacizumab vs pemetrexed disodium vs bevacizumab and pemetrexed disodium following induction therapy.

Secondary

* To determine the response rate in patients treated with these regimens.
* To evaluate the progression-free survival (PFS) of patients treated with these regimens.
* To define the toxicity of these regimens in these patients.
* To determine the frequency of polymorphisms in VEGF 3578 AA, 1154 AA, ABCB1 G2677TT/AA, and ERCC-118 TT in patients treated with induction therapy comprising paclitaxel, carboplatin and bevacizumab and determine the association between genotypes and response rate.
* To determine the association between bevacizumab and pemetrexed disodium population pharmacokinetics and patient-specific covariate with bevacizumab or pemetrexed disodium toxicity.
* To determine the frequency of TSER*3 polymorphisms in NSCLC and the association between TSER polymorphisms and benefit from pemetrexed disodium.
* To evaluate TS and ERCC1 expression by RT-PCR and MTAP mutations in existing tumor specimens as a predictor of pemetrexed disodium response.
* To evaluate polymorphisms within CYPs 2C8, 3A4, 3A5 and/or the UGT1A1 collectively or monogenically as markers for variation in efficacious and/or toxic response of individuals to treatment with taxanes.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to gender (male vs female), stage of disease (IIIB-T4Nx [with nodule in ipsilateral lung lobe and not candidate for combined chemotherapy and radiation] and IV M1a vs IV M1b vs recurrent), best response to first-time therapy (complete response/partial response vs stable disease), and smoking status (never vs smoker).

* Induction therapy (Arm I): Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Maintenance Therapy: Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Treatment begins within 6 weeks of the last day of induction chemotherapy administration.

  * Arm A: Patients receive bevacizumab IV over 30-90 minutes on day 1.
  * Arm B: Patients receive pemetrexed disodium IV over 10 minutes on day 1.
  * Arm C: Patients receive bevacizumab as in arm A and pemetrexed as in arm B. In all arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood sample collection at baseline and periodically during study for correlative studies.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 2-5 years.

ELIGIBILITY:
Inclusion Criteria (Step 1 Induction Therapy):

* Cytologically or histologically confirmed non-small cell lung cancer (NSCLC)
* Predominant non-squamous histology (NSCLC not otherwise specified allowed). Mixed tumors are categorized by the predominant cell type.
* Stage IV disease including M1a or M1b stages or recurrent disease
* Stage IIIB (T4NX) disease with ipsilateral lung lobe allowed provided patients are not candidates for combined chemotherapy or radiotherapy
* At least 12 months since prior adjuvant chemotherapy
* At least 2 weeks since prior radiotherapy
* Prior carboplatin allowed provided it was given as part of adjuvant chemotherapy
* Patients with brain metastasis must have received local therapy to the brain and have no evidence of progression in the brain for at least 2 weeks from the time of completion of local therapy, prior to registration
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Leukocytes ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ institutional upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Creatinine ≤ institutional ULN OR creatinine clearance ≥ 60 mL/min
* Urine protein:urine dipstick ≤ 0-1+ (if > 1+, urine protein creatinine ratio must be < 1)
* Measurable or non-measurable disease as defined by RECIST (Response Evaluation Criteria in Solid Tumours) criteria
* Patients with hypertension must be adequately controlled (BP < 150/100 mm Hg) with appropriate anti-hypertensive therapy or diet
* Concurrent therapeutic anti-coagulation allowed
* Fertile patients must agree to abstain from sexual intercourse or to use adequate contraceptive methods during and for at least 6 months after completion of study therapy

Exclusion Criteria (Step 1 Induction Therapy):

* Prior malignancy within the past 3 years except superficial melanoma, basal cell carcinoma, or carcinoma in situ
* Prior systemic chemotherapy for advanced stage lung cancer
* Prior use of paclitaxel, pemetrexed disodium, or bevacizumab
* Major hemoptysis within the past 4 weeks
* Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements
* History of arterial thrombotic events or major bleeding within the past 12 months
* Major surgery such as thoracotomy, laparotomy, craniotomy, or significant traumatic injury within 6 weeks prior to registration. Biopsy procedures and chest tube insertion are not considered major surgery for the purpose of this protocol.
* Core biopsy within 7 days of registration
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within the past 6 months
* Clinically significant cardiovascular disease
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* History of serious non-healing wounds, ulcers, or bone fractures
* Cavitary lesions in the lungs
* Pregnant or nursing
* Concurrent anti-retroviral therapy in patients with HIV infection

Inclusion Criteria (Step 2 Maintenance Therapy):

* Patient must have an overall stable or better response after 4 courses of induction therapy
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Patients must be registered to Step 2 within 6 weeks of the last day of chemotherapy administration on Step 1
* Acceptable bone marrow, renal and hepatic function within 2 weeks of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, MD, Study Chair — Emory University
Locations (434):
- United States (434):
  - Regional Medical Center, Anniston, Alabama
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - North Bay Cancer Center, Fairfield, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Feather River Hospital Cancer Center, Paradise, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Stanford Cancer Center, Stanford, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Kaiser Permanente at Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - North Broward Medical Center, Deerfield Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology, Pensacola, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Delnor Hospital - Geneva, Geneva, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Mitchell Memorial Cancer Center at Owensboro Medical Health System, Owensboro, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Kaiser Permanente at Woodlawn Medical Center, Baltimore, Maryland
  - Regional Cancer Center at Western Maryland Health System - Sacred Heart Campus, Cumberland, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Kaiser Permanente - Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Iris V. Henderson Cancer Center at Mercy Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Harrington Cancer Center, Amarillo, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Wheaton Franciscan Cancer Care - St. Joseph, Milwaukee, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Ramalingam SS, Dahlberg SE, Belani CP, Saltzman JN, Pennell NA, Nambudiri GS, McCann JC, Winegarden JD, Kassem MA, Mohamed MK, Rothman JM, Lyss AP, Horn L, Stinchcombe TE, Schiller JH. Pemetrexed, Bevacizumab, or the Combination As Maintenance Therapy for Advanced Nonsquamous Non-Small-Cell Lung Cancer: ECOG-ACRIN 5508. J Clin Oncol. 2019 Sep 10;37(26):2360-2367. doi: 10.1200/JCO.19.01006. Epub 2019 Jul 30. PMID 31361535
- [Derived] Wang Y, Sun Z, Sridhar A, Ramalingam SS, Wakelee HA, Gerber DE. Participation in lung cancer biospecimen studies: an analysis of the ECOG-ACRIN phase 3 E1505 and E5508 clinical trials. Lung Cancer. 2026 Feb 7;214:109304. doi: 10.1016/j.lungcan.2026.109304. Online ahead of print. PMID 41666849
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,516 patients were enrolled in the study between August 2010 and April 2015. The first patient was accrued on October 25, 2010.
Groups:
- Induction Therapy But Not Randomized to Maintenance Therapy: Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Induction Then Maintenance With Pemetrexed: Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm B receive pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
- Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm C receive bevacizumab IV over 30-90 minutes and pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
Period: Step 1: Induction Therapy
Arm/Group | Induction Therapy But Not Randomized to Maintenance Therapy | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed | Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed)
Started | 642 | 287 | 294 | 293
Completed | 65 | 287 | 294 | 293
Not Completed | 577 | 0 | 0 | 0
Not completed — Lack of Efficacy | 167 | 0 | 0 | 0
Not completed — Adverse Event | 198 | 0 | 0 | 0
Not completed — Death | 62 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 54 | 0 | 0 | 0
Not completed — Complicating disease | 13 | 0 | 0 | 0
Not completed — Alternative therapy | 12 | 0 | 0 | 0
Not completed — Symptomatic deterioration | 10 | 0 | 0 | 0
Not completed — Non-compliance | 4 | 0 | 0 | 0
Not completed — Pain | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Hospice care | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Off treatment reason not reported | 50 | 0 | 0 | 0
Period: Step 2: Maintenance Therapy
Arm/Group | Induction Therapy But Not Randomized to Maintenance Therapy | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed | Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed)
Started | 0 (Patients without complete/partial response or stable disease post induction phase weren't randomized) | 287 | 294 | 293
Completed | 0 (Patients without complete/partial response or stable disease post induction phase weren't randomized) | 1 | 0 | 1
Not Completed | 0 | 286 | 294 | 292
Not completed — Lack of Efficacy | 0 | 217 | 217 | 170
Not completed — Adverse Event | 0 | 32 | 29 | 46
Not completed — Death | 0 | 8 | 2 | 13
Not completed — Withdrawal by Subject | 0 | 11 | 21 | 27
Not completed — Alternative therapy | 0 | 2 | 4 | 5
Not completed — Other complicating disease | 0 | 2 | 5 | 9
Not completed — Symptomatic deterioration | 0 | 2 | 4 | 3
Not completed — Exceeded maximum delay in treatment | 0 | 2 | 2 | 3
Not completed — Diagnosis of progressive disease error | 0 | 1 | 1 | 0
Not completed — Financial reason | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 3 | 3
Not completed — Hospice care | 0 | 1 | 2 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 2
Not completed — Pain | 0 | 0 | 0 | 1
Not completed — Off treatment reason not reported | 0 | 4 | 4 | 10

BASELINE CHARACTERISTICS:
Population: All registered patients
Groups:
- Induction Therapy But Not Randomized: Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm C (Inductio Then Maintenance With Bevacizumab & Pemetrexed): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm C receive bevacizumab IV over 30-90 minutes and pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Induction Therapy But Not Randomized | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed) | Arm C (Inductio Then Maintenance With Bevacizumab & Pemetrexed) | Total
Number analyzed (Participants) | 642 | 287 | 294 | 293 | 1516
Age, Continuous [Median (Full Range); unit: years] | 65 [32 to 86] | 65 [43 to 85] | 63 [39 to 83] | 64 [29 to 87] | 64 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 147 | 151 | 150 | 724
  Male | 366 | 140 | 143 | 143 | 792
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 1 | 1 | 9
  Asian | 8 | 3 | 3 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 82 | 31 | 45 | 22 | 180
  White | 528 | 245 | 240 | 260 | 1273
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 18 | 5 | 4 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive.
  The primary analysis is among patients who were randomized to the maintenance therapy. Patients who received induction therapy only and did not participate in the randomization part of the study were not included in this analysis.
Time Frame: Assessed every 6 weeks during induction therapy and every 3 cycles during maintenance therapy; after discontinuation of study therapy, assessed every 3 months for 2 years and every 6 months for years 3-5
Population: All randomized patients
Measure: Median (97.5% Confidence Interval); unit: months
Arm/Group | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed | Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed)
Number analyzed (Participants) | 287 | 294 | 293
months | 14.4 [11.6 to 17.0] | 15.9 [12.7 to 20.0] | 16.4 [14.0 to 18.9]
Statistical Analysis 1: Comparison: Arm A (Induction Then Maintenance With Bevacizumab) vs Arm B (Induction Then Maintenance With Pemetrexed; Test type: Superiority; p = 0.12, Log Rank; Stratified logrank test
Statistical Analysis 2: Comparison: Arm A (Induction Then Maintenance With Bevacizumab) vs Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed); Test type: Superiority; p = 0.28, Log Rank; Stratified logrank test

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from randomization to progression or death, whichever occurs first. Progression is evaluated based on RECIST criteria and defined as appearance of one or more new lesions, unequivocal progression of existing non-target lesions, or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on current step. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  The primary analysis is among patients who were randomized to the maintenance therapy. Patients who received induction therapy only and did not participate in the randomization part of the study were not included in this analysis.
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Median (97.5% Confidence Interval); unit: months
Arm/Group | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed | Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed)
Number analyzed (Participants) | 287 | 294 | 293
months | 4.2 [3.9 to 5.0] | 5.1 [4.5 to 6.2] | 7.5 [6.6 to 9.0]

3. Secondary Outcome: Response Rate
Description: Response is evaluated based on RECIST criteria v1.1 and defined as either complete response or partial response. Complete response is defined as disappearance of all lesions. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the current step's baseline sum diameters.
  The primary analysis is among patients who were randomized to the maintenance therapy. Patients who received induction therapy only and did not participate in the randomization part of the study were not included in this analysis.
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Induction Then Maintenance With Bevacizumab) | Arm B (Induction Then Maintenance With Pemetrexed | Arm C (Induction Then Maintenance With Bevacizumab and Pemetrexed)
Number analyzed (Participants) | 287 | 294 | 293
proportion of participants | 0.125 [0.085 to 0.176] | 0.187 [0.139 to 0.244] | 0.212 [0.160 to 0.270]

4. Other Pre Specified Outcome: The Association Between Genotypes and Response Rate
Description: To determine the frequency of polymorphisms in VEGF 3578 AA, 1154 AA, ABCB1 G2677TT/AA and ERCC-118 TT in patients with NSCLC receiving paclitaxel, carboplatin and bevacizumab therapy and determine the association between genotypes and response rate.
Time Frame: as for outcome 1
Reporting Status: Not Posted

5. Other Pre Specified Outcome: The Association Between Bevacizumab and Pemetrexed Population Pharmacokinetics and Patient Specific Covariates With Bevacizumab or Pemetrexed Toxicity
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: The Frequency of TSER*3 Polymorphisms in NSCLC and the Association Between TSER Polymorphisms and Benefit From Pemetrexed
Time Frame: Assessed every 3 months for 2 years and every 6 months for years 3-5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: The Association Between TS and ERCC1 Expression and Pemetrexed Response
Time Frame: Assessed every 3 months for 2 years and every 6 months for years 3-5
Reporting Status: Not Posted

8. Other Pre Specified Outcome: The Associations Between Polymorphisms Within CYPs 2C8, 3A4, 3A5 and/or the UGT1A1 Collectively or Monogenically and Efficacy and/or Toxicities
Time Frame: Assessed every 3 months for 2 years and every 6 months for years 3-5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Description: Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Groups:
- Arm I (Induction Therapy - Carboplatin, Paclitaxel & Bevacizumab): Induction Therapy:
  Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm A (Maintenance Therapy - Bevacizumab): Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm A receive bevacizumab IV over 30-90 minutes on day 1 of every cycle until progression or unacceptable toxicity.
- Arm B (Maintenance Therapy - Pemetrexed): Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm B receive pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
- Arm C (Maintenance Therapy - Bevacizumab + Pemetrexed): Maintenance Therapy:
  Patients achieving complete response, partial response or stable disease following induction therapy are randomized to 1 of 3 treatment arms. Patients in arm C receive bevacizumab IV over 30-90 minutes and pemetrexed IV over 10 minutes on day 1 of every cycle until progression or unacceptable toxicity.
Arm/Group | Arm I (Induction Therapy - Carboplatin, Paclitaxel & Bevacizumab) | Arm A (Maintenance Therapy - Bevacizumab) | Arm B (Maintenance Therapy - Pemetrexed) | Arm C (Maintenance Therapy - Bevacizumab + Pemetrexed)
All-Cause Mortality (participants affected / at risk) | 1290/1516 | 245/287 | 240/294 | 236/293
Serious Adverse Events (participants affected / at risk) | 825/1477 | 87/284 | 107/289 | 144/286
Other Adverse Events (participants affected / at risk) | 1178/1477 | 216/284 | 222/289 | 237/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Induction Therapy - Carboplatin, Paclitaxel & Bevacizumab) (N=1477) | Arm A (Maintenance Therapy - Bevacizumab) (N=284) | Arm B (Maintenance Therapy - Pemetrexed) (N=289) | Arm C (Maintenance Therapy - Bevacizumab + Pemetrexed) (N=286)
Anemia (Blood and lymphatic system disorders) | 91 | 6 | 20 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 52 | 0 | 1 | 4
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0 | 0
Asystole (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 2 | 0 | 1 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 4 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 3 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Death NOS (General disorders) | 2 | 0 | 0 | 1
Edema face (General disorders) | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 2 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 116 | 8 | 22 | 24
Fever (General disorders) | 6 | 0 | 1 | 1
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 1
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Infusion related reaction (General disorders) | 8 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 4 | 0 | 0 | 0
Pain (General disorders) | 3 | 1 | 0 | 1
Sudden death NOS (General disorders) | 2 | 0 | 0 | 0
General and administration site - Other (General disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 7 | 0 | 0 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 8 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 32 | 0 | 5 | 5
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Esophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 15 | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 58 | 1 | 2 | 7
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 37 | 1 | 1 | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 6 | 0 | 0 | 0
Anaphylaxis (Immune system disorders) | 2 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 2 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 2 | 0 | 1 | 1
Device related infection (Infections and infestations) | 4 | 0 | 0 | 1
Duodenal infection (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Esophageal infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 24 | 1 | 6 | 6
Lymph gland infection (Infections and infestations) | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 14 | 1 | 0 | 3
Skin infection (Infections and infestations) | 2 | 0 | 3 | 1
Small intestine infection (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 3 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 0 | 2 | 3
Infections and infestations - Other (Infections and infestations) | 4 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Cardiac troponin T increased (Investigations) | 1 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 2 | 0 | 0 | 4
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 64 | 3 | 16 | 23
Neutrophil count decreased (Investigations) | 403 | 3 | 23 | 32
Platelet count decreased (Investigations) | 109 | 0 | 11 | 12
Weight gain (Investigations) | 1 | 0 | 2 | 0
Weight loss (Investigations) | 4 | 1 | 1 | 7
White blood cell decreased (Investigations) | 213 | 0 | 15 | 14
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 48 | 2 | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 42 | 1 | 5 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 16 | 0 | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 16 | 2 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 53 | 5 | 5 | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 1 | 1 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 28 | 1 | 2 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 6 | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 30 | 1 | 4 | 7
Reversible posterior leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 10 | 2 | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 0 | 0
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 3 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 2 | 5 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 8 | 12 | 1 | 8
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 161 | 47 | 13 | 54
Hypotension (Vascular disorders) | 15 | 0 | 1 | 2
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 46 | 5 | 1 | 4
Visceral arterial ischemia (Vascular disorders) | 1 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 2 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Induction Therapy - Carboplatin, Paclitaxel & Bevacizumab) (N=1477) | Arm A (Maintenance Therapy - Bevacizumab) (N=284) | Arm B (Maintenance Therapy - Pemetrexed) (N=289) | Arm C (Maintenance Therapy - Bevacizumab + Pemetrexed) (N=286)
Anemia (Blood and lymphatic system disorders) | 144 | 10 | 33 | 36
Fatigue (General disorders) | 528 | 79 | 118 | 125
Alopecia (Skin and subcutaneous tissue disorders) | 758 | 113 | 115 | 115
Constipation (Gastrointestinal disorders) | 113 | 10 | 15 | 27
Diarrhea (Gastrointestinal disorders) | 101 | 2 | 15 | 14
Mucositis oral (Gastrointestinal disorders) | 0 | 3 | 7 | 17
Nausea (Gastrointestinal disorders) | 235 | 18 | 37 | 52
Vomiting (Gastrointestinal disorders) | 93 | 3 | 14 | 21
Creatinine increased (Investigations) | 0 | 0 | 8 | 17
Lymphocyte count decreased (Investigations) | 78 | 6 | 33 | 30
Platelet count decreased (Investigations) | 93 | 0 | 0 | 0
Weight loss (Investigations) | 86 | 20 | 17 | 28
White blood cell decreased (Investigations) | 86 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 294 | 33 | 54 | 62
Dehydration (Metabolism and nutrition disorders) | 83 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 10 | 9 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 201 | 11 | 18 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 162 | 13 | 14 | 16
Dysgeusia (Nervous system disorders) | 103 | 10 | 19 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 206 | 41 | 44 | 50
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 98 | 14 | 23 | 36
Proteinuria (Renal and urinary disorders) | 0 | 41 | 2 | 39
Hypertension (Vascular disorders) | 265 | 87 | 49 | 111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT01107626/Prot_SAP_000.pdf